CLINICAL TRIAL: NCT05686135
Title: 90Second IBD for the Improvement of Self Efficacy and Quality of Life in Inflammatory Bowel Disease Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company could not update IT infrastructure to support the project
Sponsor: Jennifer Jones (Other)
Collaborators: 90 Second Health (Unknown); Takeda (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Jones, Gastroenterologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 51239
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: IBD; Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 90Second IBD (Experimental): Participants will receive 90SecondIBD weekly at no charge via text message or email linked to a website.
  Interventions: Other: 90Second IBD

INTERVENTIONS:
Other: 90Second IBD — Patients will receive 90SecondIBD weekly at no charge via text message or email linked to a website.Each 90SecondIBD letter has an attractive photo, 250 words of targeted information on a specific topic and 3 specific action suggestions on the first page. The second page is a seven-item quiz on attitudes and behavior on the designated topic. The reader gets immediate feedback and advice. The third page is a personal story of someone with IBD about this topic. Finally, there is an evaluation of the specific 90SecondIBD issue and an opportunity to recommend topics.

SUMMARY:
Patients with Inflammatory Bowel Disease (IBD) have poorer quality of life than healthy people. Despite the high prevalence of psychological issues and its profound influence on quality of life, most IBD patients have limited access to mental health support. As well, many may decline support if it is offered because mental health is often not thought of as part of IBD care. Patients may be able to access cognitive behavioural therapy (CBT) through a psychologist, however this intervention is costly and requires considerable commitment on the part of person with IBD. There is a need for new methods of reaching IBD patients to provide information on their psychological needs, and normalize the psychological effects of IBD. These new methods should integrate medical issues with psychosocial issues while being effective, scalable, and low cost to the health care system. 90SecondIBD is a novel way of delivering health information about IBD using Persuasive Design technology embedded in a planned behavior model. This project will investigate the effect of the intervention "90SecondIBD", a weekly online health letter, on IBD patients' quality of life and self efficacy. Regression modelling will be performed to explore the ability of clinical and demographic factors to predict quality of life and self efficacy scores following receipt of 90SecondIBD educational health letters weekly for 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult, resident of Canada, diagnosis of IBD, access to a computer or cell phone

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
IBD Specific Quality of life | month 0 (baseline)
  IBD specific quality of life, measured using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ). The SIBDQ comprises a total of 10 questions grouped into four domains: bowel symptoms, emotional health, systemic systems and social function. Each question is scored by a 7-point Likert scale, ranging from 1 to 7, giving an absolute score ranging from 10 (poor health related QoL) to 70 (optimal health related QoL).
IBD Specific Quality of life | month 6
  IBD specific quality of life, measured using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ). The SIBDQ comprises a total of 10 questions grouped into four domains: bowel symptoms, emotional health, systemic systems and social function. Each question is scored by a 7-point Likert scale, ranging from 1 to 7, giving an absolute score ranging from 10 (poor health related QoL) to 70 (optimal health related QoL).
IBD Specific Quality of life | month 12
  IBD specific quality of life, measured using the Short Inflammatory Bowel Disease Questionnaire (SIBDQ). The SIBDQ comprises a total of 10 questions grouped into four domains: bowel symptoms, emotional health, systemic systems and social function. Each question is scored by a 7-point Likert scale, ranging from 1 to 7, giving an absolute score ranging from 10 (poor health related QoL) to 70 (optimal health related QoL).
Self Efficacy | month 0 (baseline)
  Participant self-efficacy rating measured using the 'New General Self Efficacy Scale'. Min score: 1, max score: 8. A higher score indicates a greater self-efficacy.
Self Efficacy | month 6
  Participant self-efficacy rating measured using the 'New General Self Efficacy Scale'. Min score: 1, max score: 8. A higher score indicates a greater self-efficacy.
Self Efficacy | month 12
  Participant self-efficacy rating measured using the 'New General Self Efficacy Scale'. Min score: 1, max score: 8. A higher score indicates a greater self-efficacy.

SECONDARY OUTCOMES:
Participant Satisfaction with 90SecondIBD | month 6
  Participant Satisfaction will be assessed using 3 questions which are answered on a 1-10 point scale (no short name for the scale, is not a published measurement tool), where 1 is poor/not at all, 10 is excellent/very much : Please rate the overall value of the 90SecondIBD , Would you recommend 90SecondIBD to a friend or family member with IBD, How much did 90SecondIBD help with your management of the psychological aspects of IBD?
Participant Satisfaction with 90SecondIBD | month 12
  Participant Satisfaction will be assessed using 3 questions which are answered on a 1-10 point scale (no short name for the scale, is not a published measurement tool), where 1 is poor/not at all, 10 is excellent/very much : Please rate the overall value of the 90SecondIBD , Would you recommend 90SecondIBD to a friend or family member with IBD, How much did 90SecondIBD help with your management of the psychological aspects of IBD?

CONTACTS AND LOCATIONS:
Locations (1):
- QEII Health Sciences Centre, Halifax, N.S., Canada